CLINICAL TRIAL: NCT02627456
Title: Dose Escalating and Randomized, Placebo-Controlled, Double-Blind Study to Assess Safety, Immunogenicity, and Protective Efficacy of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites (PfSPZ Vaccine) in Healthy African Adults in Mali
Brief Title: Safety, Immunogenicity, and Protective Efficacy of Radiation Attenuated Plasmodium Falciparum NF54 Sporozoites in Healthy African Adults in Mali
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 999916004; 16-I-N004
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Malaria
Keywords: Malaria; Cryopreserved; Infection; Human; Immunization
MeSH Terms: conditions — Malaria; Infections | interventions — Saline Solution; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 1A (Experimental): (n=5), will be a safety group. Subjects will receive 1 dose of PfSPZ Vaccine (4.5x105) via DVI. All 5 subjects will receive antimalarial treatment with artesunate /amodiaquine (ASAQ) prior to PfSPZ Vaccine. Subjects will be followed for approximately 3 months post vaccination.
  Interventions: Biological: PfSPZ Vaccine; Drug: PBS and HSA Diluent; Drug: ASAQ
- 1B (Experimental): (n=S), will be a safety group. Subjects will receive 1 dose of PfSPZ Vaccine (9.0x10S) via DVI. All S subjects will receive antimalarial treatment with artesunate /amodiaquine (ASAQ) prior to PfSPZ Vaccine. Subjects will be followed for approximately 3 months post vaccination
  Interventions: Biological: PfSPZ Vaccine; Drug: PBS and HSA Diluent; Drug: ASAQ
- 1C (Experimental): (n=30), will be the targeted dose for the Pilot Safety Group. Subjects will receive 3 doses of PfSPZ Vaccine (18x105) via DVI on Day 1, 57, 113. 15 subjects will receive antimalarial treatment with artesunate /amodiaquine (ASAQ) prior to each administration of PfSPZ Vaccine, while 15 will not, except prior to PfSPZ Vaccine #3 when all 30 subjects will receive antimalarial treatment with ASAQ.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge Material; Drug: PBS and HSA Diluent; Drug: ASAQ
- 1D (Experimental): (n=15), will be the CHMI control group. Subjects will not receive any PfSPZ vaccinations but will serve as infectivity controls for CHMI. All 15 subjects will receive antimalarial treatment with ASAQ prior to PfSPZ Challenge.
  Interventions: Biological: PfSPZ Challenge Material; Drug: PBS and HSA Diluent; Drug: ASAQ
- 2 (Experimental): (n=60), will be the targeted vaccine dose arm and receive 3 doses of PfSPZ Vaccine (18x105) via DVI on Day 1, 57, 113. All subjects will receive antimalarial treatment prior to Vaccination #1 and #3 unless results obtained and analyzed from the pilot study indicate otherwise.
  Interventions: Biological: PfSPZ Vaccine; Drug: PBS and HSA Diluent; Drug: Coartem; Drug: ASAQ
- 3 (Placebo Comparator): (n=60), will be the placebo arm and receive vaccinations with normal saline via DVI on Day 1, 57, 113. All subjects will receive antimalarial treatment prior to Vaccination #1 and #3 unless results obtained and analyzed from the Pilot Study indicate otherwise.
  Interventions: Other: Normal Saline; Drug: ASAQ
- 4 (Active Comparator): (n=SS), will be group- matched (age, sex, village) controls for Arm 2 for the duration study. Subjects previously enrolled in Arm 3 may re-enroll in Arm 4. All subjects will receive antimalaria treatment at enrollment
  Interventions: Drug: Coartem

INTERVENTIONS:
Biological: PfSPZ Vaccine — PfSPZ Vaccine contains aseptic, purified, vialed, cryopreserved, radiation attenuated NF54 P. falciparum sporozoites. PfSPZ Vaccine will be delivered by DVI in the pilot and main phases of the study. Participants will receive either 1 or 3 injections.
  Arms: 1A; 1B; 1C; 2
Biological: PfSPZ Challenge Material — PfSPZ Challenge are aseptic, cryopreserved P. falciparum sporozoites used for CHMI trials. PfSPZ Challenge is not radiated, thus it is fully infections. It will be administered via DVI to participants in Arm 1c and 1d.
  Arms: 1C; 1D
Drug: PBS and HSA Diluent — The diluent for PfSPZ Vaccine and Challenge is composed of phosphate-buffered saline (PBS) and human serum albumin (HSA). Vials of sterile PBS (1.6ml) and HSA (0.5ml) will be shipped to the clinical site, where diluent composed of PBS and HSA is prepared. HSA is a licensed product which is approved for parenteral, IV administration to humans. The HSA lots are extensively tested to ensure that it is free of infectious agents as listed in the CoA and is approved for use by the Food and Drug Administration(FDA).
  Arms: 1A; 1B; 1C; 1D; 2
Other: Normal Saline — Sterile isotonic (0.9%) normal saline will be procured in the US and shipped to Mali at ambient temperature. Like the product, normal saline is a clear liquid, making it indistinguishable from the study product when drawn up into a syringe.
  Arms: 3
Drug: Coartem — Artemether/lumefantrine (coartem) is a licensed antimalarial in the US and Mali for use for uncomplicated malaria. It has an excellent safety profile and is widely used to treat malaria. Artemether /lumefantrine is a Category C pregnancy drug. Thus all female participants will undergo pregnancy testing prior to receiving this drug.
  Arms: 2; 4
Drug: ASAQ — ASAQ is a fixed dose artemisinin based combination therapy that is indicated and approved for the management of uncomplicated P. falciparum malaria. It has been shown to be as effective as artemether
  /lumefantrine when taken at a once/day dosage.
  Arms: 1A; 1B; 1C; 1D; 2; 3

SUMMARY:
Background:

Malaria is still a health problem in Sub-Saharan Africa. Death rates are stable and have even increased in some areas. There are malaria vaccines. However, researchers think repeated immunizations with a vaccine called PfSPZ may work better.

Objective:

To see if PfSPZ is safe, tolerable, and effective against malaria.

Eligibility:

Healthy adults ages 18 to 50 years who live in the Doneguebougou area in Mali

Design:

Participants will be screened with medical history and physical exam.

Participants will sign or fingerprint the consent form. They will take a survey to see how well they understand the study.

Participants will give blood and urine samples.

Participants will have at least one ECG: Soft electrodes will be stuck to the skin. A machine will record heart signals.

Participants will have HIV counseling.

Participants will be assigned to a group. Groups will get a different strength doses. Groups will get a different number of vaccines over different periods of time.

If a participant develops a rash or injection site reaction, photographs may be taken.

Participants will receive an oral anti-malaria drug during the study.

Participants will be monitored for 3 to 6 months after the last vaccine.

DETAILED DESCRIPTION:
It is known that humans can be protected against malaria by repeated immunization with radiation attenuated sporozoites. Traditionally, those sporozoites are administered by exposing the vaccinee to at least 1000 bites of sporozoite infected irradiated mosquitoes, an approach that is unsuitable for mass vaccination campaigns. Recently, Sanaria, Inc. developed a process for manufacturing, in compliance with current Good Manufacturing Practices (cGMPs) aseptic, purified, radiation attenuated cryopreserved sporozoites from a well characterized isolate of P. falciparum (Hoffman et al., 2010). This product, which is called PfSPZ Vaccine, can be administered by needle and syringe. Previous studies conducted by the Vaccine Research Center and the Navy have established that IV administration of PfSPZ Vaccine can induce sterile protection against controlled human malaria infection (CHMI) with a homologous strain of P. falciparum in up to 100% of malaria na(SqrRoot) ve individuals (Seder et al., 2013). A recent study conducted as collaboration among the Malaria Research and Training Center (MRTC, Mali), the Laboratory of Malaria Immunology and Vaccinology (LMIV) National Institute of Allergy and Infectious Diseases (NIAID), and Sanaria, Inc. (Sissoko et al., unpublished) has shown that sterile protection against naturally occurring malaria infection can be achieved, but not at the level seen in the US nor at the level desired.

The next logical step in an attempt to improve protective efficacy in the targeted endemic population is to increase the PfSPZ Vaccine dose, increasing the interval between the first and second doses to 8 weeks (as was done in WRAIR 2080 in the group receiving 3 doses of 4.5x105 PfSPZ), and reducing the numbers of doses to three. Additionally, in this study design, we also can begin to understand how the standard controlled human malaria infection (CHMI) model may be used in the field and start to explore the impact of such factors as malaria co infection and drug treatment have on vaccine responses.

The initial dose escalation pilot study will focus on safety and tolerability of the PfSPZ Vaccine. A defined number of subjects enrolled during the pilot study will also undergo further evaluation, including randomization to receive or not receive drug treatment immediately prior to each vaccination and examination of protective efficacy against homologous CHMI via PfSPZ Challenge. The targeted dose (18x105 PfSPZ Vaccine), if safe and tolerable, will be administered to a larger cohort in a double blind, randomized, placebo controlled trial to examine the protective efficacy of the vaccine against naturally occurring infection. PfSPZ Vaccinees (Arm 2) from the main study will be re enrolled the following malaria transmission along with age, sex, and village matched controls (re enrolled Arm 3, additional controls) to explore the duration of protection through another malaria transmission season.

Subjects will be recruited from rural villages in Mali. The study will be conducted as collaboration among MRTC, LMIV/NIAID, and Sanaria, Inc.

ELIGIBILITY:
* INCLUSION CRITERIA PILOT and MAIN STUDY:

Subjects must fulfill all the following criteria to be eligible for the pilot and main study:

1. Age greater than or equal to 18 and less than or equal to 50 years
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
3. In good general health and without clinically significant medical history
4. Willing to have blood samples stored for future research
5. Available for the duration of the study
6. Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to Study Day 1 to 3 months after the last vaccination.

   * Reliable methods of birth control include one of the following: confirmed pharmacologic contraceptives (parenteral) delivery; intrauterine or implantable device.
   * Reliable methods of birth control include concurrent use of a pharmacologic and a barrier method, i.e., two of the following: confirmed pharmacological contraceptives (oral, transdermal) delivery or vaginal ring AND condoms with spermicide or diaphragm with spermicide.

Non-childbearing women will also be required to report date of last menstrual period, history of surgical sterility (i.e., tubal ligation, hysterectomy) or premature ovarian insufficiency (POI), and will have urine or serum pregnancy test performed per protocol.

INCLUSION CRITERIA DURATION STUDY:

Subjects must fulfill all the following criteria to be eligible for the duration study:

1. Age greater than or equal to 18 and less than or equal to 52 years
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
3. In good general health and without clinically significant medical history
4. Willing to have blood samples stored for future research
5. Available for the duration of the study
6. Participated in the main phase of this protocol (Arms 2,3) AND received all three vaccinations OR suitable to serve as a matched control for such an individual.

EXCLUSION CRITERIA PILOT and MAIN STUDY:

A subject will be excluded from participating in the pilot or main trial if any one of the following criteria is fulfilled:

1. Pregnancy, as determined by a positive urine or serum human choriogonadotropin (beta-hCG) test (if female)
2. Currently breast-feeding (if female)
3. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
4. Hemoglobin, WBC, absolute neutrophils, and platelets outside the local laboratory defined limits of normal (subjects may be included at the investigator's discretion for not clinically significant values)
5. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal (subjects may be included at the investigator's discretion for not clinically significant values)
6. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B (HBV)
7. Known or documented sickle cell disease by history (Note: known sickle cell trait is NOT exclusionary)
8. Clinically significant abnormal ECG
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
10. History of receiving any investigational product within the past 30 days
11. Participation or planned participation in a clinical trial with an investigational product prior to completion of the follow-up visit 28 days following last vaccination OR planned participation in an investigational vaccine study until the last required protocol visit
12. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
13. History of a severe allergic reaction or anaphylaxis
14. Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has rquired the use of oral or parenteral corticosteroids at any time during the past 2 years.
15. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia
16. Known immunodeficiency syndrome
17. Known asplenia or functional asplenia
18. Use of:

    * Chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of vaccination
    * Use of antimalarials or systemic antibiotics with known antimalarial activity within 30 days prior to the first vaccine
19. Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to Vaccination #1 and every subsequent vaccination day
20. Receipt of immunoglobulins and/or blood products within the past 6 months
21. Previous receipt of an investigational malaria vaccine in the last 5 years
22. Known allergies or contraindication against: ASAQ or Coartem
23. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

EXCLUSION CRITERIA DURATION STUDY:

Subjects must

1. Known to be pregnant by history or as determined by a positive urine or serum human choriogonadotropin (Beta-hCG) test (if female)
2. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and comply with the study protocol
3. Hemoglobin, WBC, absolute neutrophils, and platelets outside the local laboratory defined limits of normal (subjects may be included at the investigator's discretion for not clinically significant values)
4. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal (subjects may be included at the investigator's discretion for not clinically significant values)
5. Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B (HBV)
6. Known or documented sickle cell disease by history (Note: known sickle cell trait is NOT exclusionary)
7. Receipt of artemether/lumefantrine within less than 14 days from enrollment.
8. Knwn allergies or contraindications (such as significant cardiac disease; prolonged QTc greater than 450 ms; currently taking medications that may prolong your QTc; serious side effects from artemether/lumefantrine in the past) to study treatment (artemether/lumefantrine)
9. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis
10. Enrollment in another investigational trial during the study period (participating in screening for other investigational trials is permitted).
11. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
12. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sj(SqrRoot)(Delta)gren s syndrome, or autoimmune thrombocytopenia
13. Known immunodeficiency syndrome
14. Known asplenia or functional asplenia
15. Use of Chronic (greater than or equal to 14 days) oral or intravenous corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of Study Day 0
16. Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a participant participating in the trial, interfere with the evaluation of the study objectives, or would render the subject unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 409 (Actual)
Dates: Start 2015-12-09; Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-03 (Actual)

PRIMARY OUTCOMES:
Duration | For 24 weeks starting approximately 1 year post vaccination #3
  P. falciparum blood stage infection defined as time to first positive blood smear (detection of at least 2 P. falciparum parasites by microscopic examination of 0.5 muL)
Safety | Approximately within 7 days after each vaccination and SAEs related to vaccination
  Measure the incidence and severity of local and systemic adverse events occurring within 7 days after each vaccine administration and SAE related to vaccination.

SECONDARY OUTCOMES:
Protective Efficacy (pilot phase) | Immediately following PfSPZ CHMI
  P. falciparum blood stage infection defined as detection of at least 2 P. falciparum parasites by microscopic examination of 0.5 (Micro)L starting immediately following PfSPZ CHMI(Arms lc, ld)
Protective Efficacy (main phase) | Immediately following 3rd vaccination
  P. falciparum blood stage infection defined as detection of at least 2 P. falciparum parasites by microscopic examination of 0.5 muL starting immediately following Vaccination #3 (Arms 2, 3)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- University of Bamako (USTTB/MRTC), Bamako, Mali

REFERENCES:
- [Background] Hoffman SL, Billingsley PF, James E, Richman A, Loyevsky M, Li T, Chakravarty S, Gunasekera A, Chattopadhyay R, Li M, Stafford R, Ahumada A, Epstein JE, Sedegah M, Reyes S, Richie TL, Lyke KE, Edelman R, Laurens MB, Plowe CV, Sim BK. Development of a metabolically active, non-replicating sporozoite vaccine to prevent Plasmodium falciparum malaria. Hum Vaccin. 2010 Jan;6(1):97-106. doi: 10.4161/hv.6.1.10396. Epub 2010 Jan 21. PMID 19946222
- [Background] Mordmuller B, Supan C, Sim KL, Gomez-Perez GP, Ospina Salazar CL, Held J, Bolte S, Esen M, Tschan S, Joanny F, Lamsfus Calle C, Lohr SJ, Lalremruata A, Gunasekera A, James ER, Billingsley PF, Richman A, Chakravarty S, Legarda A, Munoz J, Antonijoan RM, Ballester MR, Hoffman SL, Alonso PL, Kremsner PG. Direct venous inoculation of Plasmodium falciparum sporozoites for controlled human malaria infection: a dose-finding trial in two centres. Malar J. 2015 Mar 18;14:117. doi: 10.1186/s12936-015-0628-0. PMID 25889522
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Derived] Sissoko MS, Healy SA, Katile A, Zaidi I, Hu Z, Kamate B, Samake Y, Sissoko K, Mwakingwe-Omari A, Lane J, Imeru A, Mohan R, Thera I, Guindo CO, Dolo A, Niare K, Koita F, Niangaly A, Rausch KM, Zeguime A, Guindo MA, Bah A, Abebe Y, James ER, Manoj A, Murshedkar T, Kc N, Sim BKL, Billingsley PF, Richie TL, Hoffman SL, Doumbo O, Duffy PE. Safety and efficacy of a three-dose regimen of Plasmodium falciparum sporozoite vaccine in adults during an intense malaria transmission season in Mali: a randomised, controlled phase 1 trial. Lancet Infect Dis. 2022 Mar;22(3):377-389. doi: 10.1016/S1473-3099(21)00332-7. Epub 2021 Nov 18. PMID 34801112